CLINICAL TRIAL: NCT05713877
Title: DELIRE-ICU: A Randomised Controlled Feasibility Trial of Melatonin vs Placebo in the Treatment of Delirium in the Intensive Care Unit
Brief Title: Melatonin for Treatment of Delirium in Critically Ill Adult Patients
Acronym: DELIRE-ICU
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-3247
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Delirium
Keywords: Melatonin; Intensive care; Feasibility; Treatment; Critically ill; ICU
MeSH Terms: conditions — Delirium; Critical Illness | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All study personnel, care provider, patients and their families will remain blinded. Randomization will be performed by members of the Pharmacy Research Department.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Enteral melatonin 9 mg (Experimental): Melatonin 9 mg from a 1 mg/mL oral suspension of melatonin in ORA-BLEND SF® (sugar-free flavoured suspending vehicle). Final volume in the oral syringe will be 9 mL.
  Interventions: Drug: Melatonin
- Enteral placebo (Placebo Comparator): ORA-BLEND SF® (sugar-free flavoured suspending vehicle). Final volume in the oral syringe will be 9 mL.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — Study drug will be given at 21:00 daily, starting on the day of enrolment until delirium resolution, hospital discharge, death, or up to 14 days. The study medication will be given by mouth (PO or per os) or, if needed, via the feeding tube.
  Arms: Enteral melatonin 9 mg
Drug: Placebo — Study drug will be given at 21:00 daily, starting on the day of enrolment until delirium resolution, hospital discharge, death, or up to 14 days. The study medication will be given by mouth (PO or per os) or, if needed, via the feeding tube.
  Arms: Enteral placebo

SUMMARY:
The purpose of this study is to determine the feasibility of conducting a randomized controlled trial (RCT) with melatonin for treatment of delirium in critically ill adult patients. From a feasibility perspective, the investigators believe that the proposed design will achieve the minimum enrollment rate necessary to conduct a future RCT on a larger scale.

DETAILED DESCRIPTION:
The prevalence of delirium is high in the intensive care unit (ICU), yet there is no pharmacological treatment that has been proven effective. The investigators hypothesize that melatonin, given on a daily basis at 21:00, will safely decrease the mean duration of a delirium episode in ICU patients. The current literature evaluating melatonin as a treatment for delirium is lacking, therefore more studies are needed.

It is estimated that an alteration of sleep pattern can be found in up to 75% of patients with delirium. This raises the hypothesis that prevention and treatment of sleep disorders could potentially improve delirium. Sleep and circadian rhythm disturbances are associated with low endogenous melatonin secretion and studies have shown that it also occurs in patients with delirium.

Thus, the objective is to conduct a phase II double blind, placebo-controlled randomized trial comparing melatonin 9 mg to placebo to evaluate the feasibility of a future large-scale RCT. Participants will be followed during their stay in the ICU and after their transfer on another unit up to a maximum of 14 days. Feasibility of the larger trial will mainly be based on enrollment rates.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older admitted to the intensive care unit;
* Anticipated ICU stay > 48 hours;
* ICDSC score greater than or equal to 4 for a maximum of 48 hours prior to randomization.

Exclusion Criteria:

* Known allergy or hypersensitivity to melatonin or to ingredients in ORA-BLEND SF®;
* Use of melatonin within 24 hours prior to randomization;
* Presence of severe structural brain injury (intracranial hemorrhage or traumatic brain injury), severe major neurocognitive disorder, advanced neurodegenerative disease or hepatic encephalopathy;
* Diagnosis of schizophrenia, bipolar affective disorder, psychotic depression, uremic encephalopathy or alcohol withdrawal;
* Presence of active seizures, coma, aphasia or severe intellectual disability;
* Limited short-term vital prognosis;
* Diagnosis of delirium prior to ICU admission;
* Pregnancy or breastfeeding;
* Absolute contraindication to receive enteral medication;
* Inability to understand or speak English or French;
* Total blindness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Enrollment rate | 8 months
  Average enrollment rate of participants per month.
Clinical: Duration of delirium | 14 days
  Compare the average duration of an episode of delirium defined as the number of days with ICDSC score ≥4 between the 2 groups.

SECONDARY OUTCOMES:
Feasibility: Study adherence | 8 months
  Proportion of administered doses in the prescribed dose administration window (between 19:00 and 23:00 hours) divided by total number of eligible study days.
Feasibility: Consent rate | 8 months
  Proportion of participants recruited among eligible patients.
Clinical: Adverse events | 14 days
  Incidence of adverse events reported in the Canadian melatonin monograph (i.e. headache and nausea) observed by the investigators or reported by the treating team.

OTHER OUTCOMES:
Feasibility: Completion of study | 8 months
  Proportion of participants who completed the study and reasons associated with withdrawal.
Feasibility: MDAS assessment time (minutes) | 8 months
  Time required for the administration of the Memorial Delirium Assessment Scale (MDAS).
  Values from 0 to 30. A higher score means a worse outcome.
Feasibility: Completion of ICDSC | 8 months
  Proportion of missing data in the completion of the Intensive Care Delirium Screening Checklist (ICDSC).
  Values from 0 to 8. A higher score means a worse outcome.
Clinical: Antipsychotics dose (mg) administered to participants | 14 days
  Cumulative dose of de novo antipsychotics, reported in haloperidol equivalent dose, received by participants during delirium.

CONTACTS AND LOCATIONS:
Overall Officials: François Marquis, M.D., M.A., Principal Investigator — Centre intégré universitaire de santé et de services sociaux (CIUSSS) de l'Est-de-l'Île-de-Montréal
Locations (1):
- Hopital Maisonneuve-Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flacker JM, Lipsitz LA. Neural mechanisms of delirium: current hypotheses and evolving concepts. J Gerontol A Biol Sci Med Sci. 1999 Jun;54(6):B239-46. doi: 10.1093/gerona/54.6.b239. PMID 10411009
- [Background] Pandharipande PP, Morandi A, Adams JR, Girard TD, Thompson JL, Shintani AK, Ely EW. Plasma tryptophan and tyrosine levels are independent risk factors for delirium in critically ill patients. Intensive Care Med. 2009 Nov;35(11):1886-92. doi: 10.1007/s00134-009-1573-6. Epub 2009 Jul 9. PMID 19588122
- [Background] Stollings JL, Kotfis K, Chanques G, Pun BT, Pandharipande PP, Ely EW. Delirium in critical illness: clinical manifestations, outcomes, and management. Intensive Care Med. 2021 Oct;47(10):1089-1103. doi: 10.1007/s00134-021-06503-1. Epub 2021 Aug 16. PMID 34401939
- [Background] Sun T, Sun Y, Huang X, Liu J, Yang J, Zhang K, Kong G, Han F, Hao D, Wang X. Sleep and circadian rhythm disturbances in intensive care unit (ICU)-acquired delirium: a case-control study. J Int Med Res. 2021 Mar;49(3):300060521990502. doi: 10.1177/0300060521990502. PMID 33730927
- [Background] Weinhouse GL, Schwab RJ, Watson PL, Patil N, Vaccaro B, Pandharipande P, Ely EW. Bench-to-bedside review: delirium in ICU patients - importance of sleep deprivation. Crit Care. 2009;13(6):234. doi: 10.1186/cc8131. Epub 2009 Dec 7. PMID 20053301
- [Background] Farasat S, Dorsch JJ, Pearce AK, Moore AA, Martin JL, Malhotra A, Kamdar BB. Sleep and Delirium in Older Adults. Curr Sleep Med Rep. 2020;6(3):136-148. doi: 10.1007/s40675-020-00174-y. Epub 2020 Jul 27. PMID 32837850
- [Background] Burry L, Scales D, Williamson D, Foster J, Mehta S, Guenette M, Fan E, Detsky M, Azad A, Bernard F, Rose L. Feasibility of melatonin for prevention of delirium in critically ill patients: a protocol for a multicentre, randomised, placebo-controlled study. BMJ Open. 2017 Mar 30;7(3):e015420. doi: 10.1136/bmjopen-2016-015420. PMID 28363933
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272